CLINICAL TRIAL: NCT03116074
Title: Interactive Patient-Centered Discharge Toolkit to Promote Self-Management During Transitions (PDTK) & PREventing Adverse Events Post-Discharge Through Proactive Identification, Multidisciplinary Communication, and Technology (PREDICT)
Brief Title: Interactive Digital Health Tools to Improve Patient Safety in Acute Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Crico (Other)
Responsible Party: Principal Investigator, Anuj K. Dalal, MD, Associated Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016P001137
Record Dates: First submitted 2017-03-29; First posted 2017-04-14 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Transitions of Care; Patient Portals; General Medicine; Discharge Checklist; Patient-provider Communication; Adverse Event; Readmission

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Study 1: Pre-intervention 1 (No Intervention): Usual care.
  Patients/caregivers do not have access to patient portal. Providers have access to safety dashboard without discharge preparation indicator. Providers do not have access to secure patient-provider messaging tools.
- Study 1: Post-intervention (Experimental): Patient-Centered Discharge Toolkit: patient portal and provider safety dashboard PLUS patient pre-discharge checklist, provider discharge preparation indicator, secure patient-provider messaging
  Patients/caregivers have access to patient portal with discharge module (pre-discharge preparation checklist) and secure patient-provider messaging tools activated. Providers have access to discharge preparation indicator on safety dashboard and secure patient-provider messaging tools.
  Interventions: Behavioral: Interactive Digital Health Tools
- Study 1: Pre-intervention 2 (No Intervention): Usual care PLUS patient portal and provider safety dashboard.
  Patients/caregivers have access to patient portal but not discharge module or secure patient-provider messaging tools. Providers have access to safety dashboard without discharge preparation indicator. Providers do not have access to secure patient-provider messaging tools.
- Study 2: Pre-intervention (No Intervention): Usual care on three general medicine units.
  Patients/caregivers do not have access to the discharge preparation checklist. Providers do not have access to the safety dashboard.
- Study 2: Post-intervention (Experimental): Patients/caregivers have access to the discharge preparation checklist. Providers have access to safety dashboard.
  Interventions: Behavioral: Interactive Digital Health Tools

INTERVENTIONS:
Behavioral: Interactive Digital Health Tools — Discharge checklist, discharge video, safety dashboard enhanced with discharge preparation indicator, secure patient-provider messaging, condition-specific educational videos
  Arms: Study 1: Post-intervention; Study 2: Post-intervention

SUMMARY:
Study 1: The goal of this study is to implement and evaluate an interactive patient-centered discharge toolkit (PDTK) to engage patients and care partners in discharge preparation and communication with providers after discharge. The aims of this study are to:

1. To refine and implement an interactive PDTK on a general medicine unit that patient and caregivers can use to prepare for discharge and communicate with key providers during the transition home.
2. To evaluate the impact of the PDTK on patient activation (primary outcome). Patient reported self-efficacy after discharge; post-discharge healthcare resource utilization; and perception of patient-provider communication will be measured as secondary outcomes.
3. To identify barriers and facilitators of implementation, adoption, and use of the PDTK by patients, caregivers, and providers using qualitative and quantitative methods.

Study 2: The goal of this study is to expand the use of previously developed patient safety dashboards and patient-centered discharge checklists to three general medicine units in an affiliated community hospital. The safety dashboard and interactive pre-discharge checklist are cognitive aids for clinicians and patients, respectively, that serve to facilitate early detection of patients at risk for preventable harm, including suboptimal discharge preparation. The aims of this study are to:

1. Enhance the safety dashboard and interactive pre-discharge checklist to include "smart" notifications for hospital-based clinicians when patients are at high risk for adverse events or have identified specific concerns related to discharge based on their checklist responses.
2. Expand intervention to general medical units at our community hospital-affiliate, BWFH.
3. Evaluate impact on post-discharge AEs for patients discharged from BWFH who are at risk for preventable harm and hospital readmission.

DETAILED DESCRIPTION:
Study 1: The transition from the hospital is a vulnerable time for patients and stressful for caregivers-new treatments have been initiated, conditions require close monitoring, and the plan of care is in flux. Achieving a high-quality transition requires effective understanding of the discharge plan by patients/caregivers as well as seamless communication with key inpatient providers to address patients' concerns during and immediately after hospitalization. We designed an interactive patient-centered discharge toolkit (PDTK) that is accessible from an acute care patient portal. The PDTK allows patients and/or caregivers to self-assess discharge preparedness via a validated, pre-discharge checklist tool and communicate directly with key members of the care team. Information entered by the patient regarding their discharge preparedness is presented to the unit-based care team on an interactive safety dashboard so that providers can address any barriers prior to discharge. After discharge, patients can communicate directly with providers about issues or concerns that arise prior to follow-up with their ambulatory providers.

The PDTK will be implemented and evaluated for patients admitted to and discharged from general medicine units. The RE-AIM (reach, effectiveness, adoption, implementation, and maintenance) framework will be used to inform research questions and methods that guide implementation and evaluation. A pre-post study will be performed in which the primary outcome is analyzed as the proportion of patients with Patient Activation Measure (PAM) Levels 3 or 4 at discharge. Approximately 358 patients will be enrolled to provide adequate power to detect an improvement in the primary outcome from 72% to 84%. Quantitative and qualitative methods will be used to assess implementation, adoption, and use of the intervention.

Study 2: Our project proposes to address gaps in functionality of commercially available EHR systems through evaluation of novel, EHR-integrated HIT tools. We previously designed, developed, and implemented the patient safety dashboard and interactive pre-discharge checklist to engage clinicians and patients in systematically addressing safety threats in each of several domains. By integrating clinical data of several different types, these tools serve to reduce cognitive load and improve decision-making for clinicians. In this way, these tools represent a preventative intervention that mitigates risk in each domain by suggesting corrective action corresponding to institutional safety guidelines.

Studying the effectiveness of these tools on post-discharge outcomes will improve knowledge, technical capability, and clinical practice related to patient safety during transitions of care. Specifically, our project will advance scientific knowledge by quantifying the post-discharge impact of an intervention that changes clinical practice by enabling hospital-based clinicians to proactively institute corrective action for "at risk" patients who may require additional surveillance and supportive services during transitions. Also, we will establish the technical feasibility of spreading customized, third-party digital health applications that fill critical safety gaps in commercially available EHRs; expanding to a community hospital has clear implications for adoption and validation of this technology in different practice settings.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, >18 years of age, English-speaking
* Caregivers >18 years of age designated by patient or patient's healthcare proxy
* Male or female healthcare providers of enrolled patients

Exclusion Criteria:

-Non-English speaking patients for whom we cannot identify an English-speaking healthcare proxy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Study 1: Patient or Caregiver Activation at Discharge | 16 months
  The short version of the Patient Activation Measure (PAM®) or Caregiver Activation Measure (CAM®) tool will be administered to all enrolled patients or enrolled patient's designated caregivers at discharge.
Study 2: Potential Post-Discharge Adverse Events | 24 months
  Potential post-discharge adverse events will be measured as the number of new or worsening symptoms or signs per patient

SECONDARY OUTCOMES:
Study 1: Patient Reported Self-Efficacy | 16 months
  Patients or designated caregivers will be asked at 30 days after discharge to rate the degree of involvement (5-point Likert scale) in their discharge plan in each of four domains: executing the discharge plan of care; taking discharge medications; self-managing conditions; adhering to the follow-up plan
Study 1: Patient or Caregiver Activation at 30-days Post-Discharge | 16 months
  The short version of the Patient Activation Measure (PAM®) or Caregiver Activation Measure (CAM®) tool will be administered to all enrolled patients or enrolled patient's designated caregivers at 30-days after discharge
Study 1: Healthcare Resource Utilization | 16 months
  Healthcare resource utilization will be measured as the aggregate number of ambulatory clinic visits (PCPs, specialists), emergency department visits, and hospital re-admissions during the 30-day post-discharge period via hospital administrative databases and by asking patients/caregivers about utilization of resources outside our healthcare network on a 30-day post-discharge phone call.
Study 1: Provider perceptions of patients' discharge preparedness and patient-provider communication regarding the discharge process | 16 months
  Assessed using surveys (5-point Likert scale) administered to patients' providers (nurse, attending, residents, physician assistants) at discharge.
Study 1: Patient perceptions of their discharge preparedness and patient-provider communication regarding the discharge process during hospitalization and the post-discharge transition period. | 16 months
  Assessed using surveys (5-point Likert scale) administered to patients/caregivers at discharge, and during the 30-day patient phone call.
Study 2: Actual Post-Discharge Adverse Events | 24 months
  Actual post-discharge adverse events will be measured as the number of adverse events per patient
Study 2: Preventable Post-Discharge Adverse Events | 24 months
  Actual post-discharge adverse events related to preventable harm will be measured as the number of post-discharge adverse events per patient related to a specific safety risk domain identified during index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Anuj K Dalal, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dalal AK, Piniella N, Fuller TE, Pong D, Pardo M, Bessa N, Yoon C, Lipsitz S, Schnipper JL. Evaluation of electronic health record-integrated digital health tools to engage hospitalized patients in discharge preparation. J Am Med Inform Assoc. 2021 Mar 18;28(4):704-712. doi: 10.1093/jamia/ocaa321. PMID 33463681
- [Derived] Fuller TE, Pong DD, Piniella N, Pardo M, Bessa N, Yoon C, Boxer RB, Schnipper JL, Dalal AK. Interactive Digital Health Tools to Engage Patients and Caregivers in Discharge Preparation: Implementation Study. J Med Internet Res. 2020 Apr 28;22(4):e15573. doi: 10.2196/15573. PMID 32343248
- See also: AHRQ Project Site — https://healthit.ahrq.gov/ahrq-funded-projects/interactive-patient-centered-discharge-toolkit-promote-self-management-during